CLINICAL TRIAL: NCT00156039
Title: A Randomized Trial of Follow-up Strategies in Breast Cancer
Brief Title: Randomized Trial of Follow-up Strategies in Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Breast Cancer Initiative (Unknown)
Responsible Party: Dr. Eva Grunfeld, Cancer Outcomes Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OCOG-1997-FUP; CBCRI-grant-010413
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Follow-up Strategy; Follow-up Care; Family Physician; Oncologist
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Follow-up Strategy for Breast Cancer

SUMMARY:
The purpose of this study is to determine whether family physician 'routine follow-up care' of women with breast cancer in remission is an acceptable alternative to the existing system of specialist follow-up. Primary outcome measure are event rates of oncological catastrophes and quality of life.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer on well follow-up at regional cancer centres in Ontario and Manitoba
* Diagnosed at least 12 months previously (range 9-15 months)
* Without evidence of active disease (i.e., stages IIIB and IV excluded)
* Free from any primary treatment complications

Exclusion Criteria:

* Primary treatment at least 3 months previously, except for continued use of tamoxifen
* Still experiencing complications of primary treatment (patients will become eligible once complications resolve provided they are within the 6 month window)
* Unable to identify an acceptable family physician to provide follow-up
* Language or literacy skills inconsistent with completing questionnaires
* Unable to comply with study protocol including completion of questionnaires
* Previously enrolled in a study which requires continued follow-up in specialist or peripheral clinics
* Actively followed at a cancer centre for another primary cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 968 (Actual)
Dates: Start 1997-01; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Rate of clinically catastrophic events | Up to 5 yrs after randomization
Rate of Karnofsky performance status < 70 | Up to 5 yrs after randomization
Psychosocial well being of patients in remission | Up to 5 yrs after randomization

SECONDARY OUTCOMES:
Health Related Quality of Life after recurrence | Up to 5 yrs after randomization
Survival | Up to 5 yrs after randomization
Economic evaluation | Up to 5 yrs after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Eva Grunfeld, MD, Study Chair — Cancer Care Nova Scotia; Mark Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (5):
- Canada (5):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Ottawa Hospital - Integrate Cancer Program, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario

REFERENCES:
- [Result] Grunfeld E, Levine MN, Julian JA, Coyle D, Szechtman B, Mirsky D, Verma S, Dent S, Sawka C, Pritchard KI, Ginsburg D, Wood M, Whelan T. Randomized trial of long-term follow-up for early-stage breast cancer: a comparison of family physician versus specialist care. J Clin Oncol. 2006 Feb 20;24(6):848-55. doi: 10.1200/JCO.2005.03.2235. Epub 2006 Jan 17. PMID 16418496